CLINICAL TRIAL: NCT05243979
Title: The Relation Between Thyroid , Parathyroid Hormones and Estimated Glomerular Filtration Rate in Chronic Kidney Disease Patients in Assiut
Brief Title: The Relation Between Thyroid , Parathyroid Hormones and eGFR in CKD Patients in Assiut
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Magdy Ahmed Mohammed, Resident doctor, Assiut University
Other Study IDs: Thyroid, Parathyroid CKD
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Thyroid; Parathyroid Diseases; CKD
Keywords: Thyroid; Parathyroid Diseases; CKD
MeSH Terms: conditions — Thyroid Diseases; Parathyroid Diseases | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group (A): 40 patients with CKD (1-3) not on renal replacement therapy.
  Interventions: Radiation: DEXA scan
- Group (B): 40 persons with normal kidney function and GFR ( control ).

INTERVENTIONS:
Radiation: DEXA scan — bone study
  Groups: Group (A)

SUMMARY:
To evaluate the relation between thyroid, parathyroid hormones and estimated glomerular filtration rate in chronic kidney disease .

DETAILED DESCRIPTION:
CKD is defined as abnormalities of kidney structure or function, present for >3 months, with implications for health. CKD is classified based on Cause, GFR category (G1-G5), and Albuminuria category (A1-A3) .

The global prevalence of CKD is 13.4%, with 10.6% being stages 3-5 ,Over the past 10 years, the death rate due to CKD has increased by 31.7% .

CKD patients remain sometimes asymptomatic, presenting the complications typical of renal dysfunction only in more advanced stages. Its treatment can be conservative usually in patients with glomerular filtration rate above 15 ml/minute without indications of dialysis or replacement therapy .

In CKD patients the changes of endocrine system levels may arise from several causes as the kidney is the site of degradation & synthesis of many different hormones .

So thyroid and parathyroid hormones dysfunction has been recognized as common co-morbidity that is often diagnosed with CKD .

Thyroid hormone is one of the most important hormones in the human body as it regulates majority of the body's physiological actions .

Parathyroid hormone (PTH) is one of the most important hormones required for the maintenance of calcium and phosphate homeostasis .

Chronic kidney disease metabolic bone disorder (CKD-MBD) among patients with end stage renal disease ranges from 33% to 67%, and its severity tends to increase with the progression of the kidney damage & high mortality rates .

CKD-MBD causes bone abnormalities that affect turnover, volume, mineralization, vascular, linear growth, and density, and soft tissue calcification .

ELIGIBILITY:
Inclusion Criteria:

* 1. CKD patients 2. Age (18-80 years) 3. Diabetic nephropathy 4. Hypertensive nephropathy 5. Chronic pyelonephritis 6. Obstructive nephropathy 7. Polycystic kidney 8. Gout nephropathy 9. Nephrosclerosis

Exclusion Criteria:

* 1. Patients underage of 18 and above 80 2. Patients with history of thyroidectomy and parathyroidectomy 3. Patients with history of thyroid and parathyroid disease before diagnosis of CKD 4. Malignancy

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Assuit University Hospital -Internal medicine department (Inpatient and outpatient settings).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
The Relation between thyroid , parathyroid hormones and estimated glomerular filtration rate in chronic kidney disease patients in Assiut | Baseline
  To evaluate the relation between thyroid, parathyroid hormones and estimated glomerular filtration rate in chronic kidney disease different stages

CONTACTS AND LOCATIONS:
Overall Officials: Sara Magdy, Study Chair — Assiut University; Hanan Mahmoud, Study Chair — Assiut University; Nashwa Mostafa, Study Chair — Assiut University

REFERENCES:
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) Diabetes Work Group. KDIGO 2020 Clinical Practice Guideline for Diabetes Management in Chronic Kidney Disease. Kidney Int. 2020 Oct;98(4S):S1-S115. doi: 10.1016/j.kint.2020.06.019. No abstract available. PMID 32998798
- [Background] Laible M, Horstmann S, Rizos T, Rauch G, Zorn M, Veltkamp R. Prevalence of renal dysfunction in ischaemic stroke and transient ischaemic attack patients with or without atrial fibrillation. Eur J Neurol. 2015 Jan;22(1):64-9, e4-5. doi: 10.1111/ene.12528. Epub 2014 Aug 4. PMID 25091540
- [Background] Banerjee D, Jha V. Vitamin D and Cardiovascular Complications of CKD: What's Next? Clin J Am Soc Nephrol. 2019 Jun 7;14(6):932-934. doi: 10.2215/CJN.12581018. Epub 2019 May 7. No abstract available. PMID 31064752
- [Background] Ammirati AL. Chronic Kidney Disease. Rev Assoc Med Bras (1992). 2020 Jan 13;66Suppl 1(Suppl 1):s03-s09. doi: 10.1590/1806-9282.66.S1.3. PMID 31939529
- [Background] Kuczera P, Adamczak M, Wiecek A. Endocrine Abnormalities in Patients with Chronic Kidney Disease. Pril (Makedon Akad Nauk Umet Odd Med Nauki). 2015;36(2):109-18. doi: 10.1515/prilozi-2015-0059. PMID 27442377
- [Background] Peters J, Roumeliotis S, Mertens PR, Liakopoulos V. Thyroid hormone status in patients with impaired kidney function. Int Urol Nephrol. 2021 Nov;53(11):2349-2358. doi: 10.1007/s11255-021-02800-2. Epub 2021 Mar 8. PMID 33682051
- [Background] Guo Y, Wang Q, Lu C, Fan P, Li J, Luo X, Chen D. New parathyroid function index for the differentiation of primary and secondary hyperparathyroidism: a case-control study. BMC Endocr Disord. 2020 Jan 8;20(1):5. doi: 10.1186/s12902-019-0487-8. PMID 31914999
- [Background] Habas E Sr, Eledrisi M, Khan F, Elzouki AY. Secondary Hyperparathyroidism in Chronic Kidney Disease: Pathophysiology and Management. Cureus. 2021 Jul 14;13(7):e16388. doi: 10.7759/cureus.16388. eCollection 2021 Jul. PMID 34408941